CLINICAL TRIAL: NCT05571241
Title: Accelerated vs Traditional Rehabilitation Protocol Following Ligament Reconstruction Tendon Interposition Surgery Using Interference Screw Fixation for 1st CMC Arthritis .
Brief Title: Ligament Reconstruction in an Accelerated Rehabilitation Protocol
Status: Withdrawn | Type: Observational
Why Stopped: No resident involvement
Sponsor: Dr. David Pichora (Other)
Responsible Party: Sponsor-Investigator, Dr. David Pichora, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Other Study IDs: SURG-288-14
Record Dates: First submitted 2014-04-24; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fast rehabilitation program: conventional rehabilitation
  Interventions: Behavioral: Fast rehabilitation program

INTERVENTIONS:
Behavioral: Fast rehabilitation program — 1-2 weeks (first post-op visit): Long thumb spica splint removed; Staples/stitches removed; Short hand-based thumb spica fitted for the patient Start Active Range of Motion Exercises (AROM) for thumb Add active assisted rang of motion exercises (AAROM) if no significant progress 6 weeks: Gradually wean off of splint during the day; wear for protection and/or more strenuous daily activities 6-8 weeks: Passive Range of Motion Exercises (PROM) (ie. stretching), if needed - (ie. No significant changes in ROM of thumb) 8-10 weeks: Resisted exercises/activities without splint on

SUMMARY:
The investigators have found that their patients who get earlier rehabilitation following ligament reconstruction and tendon interposition (LRTI) surgery with interference screws have experienced better outcomes. The investigators hypothesis is that when formally comparing these patients who are exposed to the rehabilitation protocol earlier compared to later, the investigators will see statistically better outcomes.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the 1st carpometacarpal (CMC) joint is a significant cause of hand pain, dysfunction, disability, and visible deformity. Surgery in the form of ligament reconstruction and tendon interposition (LRTI)is often indicated when less invasive procedures fail. Following LRTI procedures, the accepted classic protocol throughout the literature has been to place patients in a thumb-immobilizing spica cast or splint for 4-6 weeks and then begin rehabilitation exercises. Following this, a gradual progressive rehabilitation protocol is initiated which usually focuses on thumb range of motion, pinch strength, and hand function. This standard form of rehabilitation has shown improvements in pain, function, and satisfaction. However, because these patients are usually kept immobilized until 4-6 weeks post-operatively in order for the tendon graft to incorporate and become stable, stiffness can develop in the thumb as a result. This leads to more time off work and without full and unrestricted use of the hand. Due to their higher pullout strength compared to conventional tendon fixation, the use of interference screws in LRTI procedures may allow for earlier initiation of a more accelerated rehabilitation protocol compared to the standard 4-6 weeks of immobilization prior to rehabilitation. Over the past year at the investigators center the investigators have begun post-operative mobilization and rehabilitation on the first post-op visit at 10-14 days following LRTI with the use of an interference screw. Anecdotally, the investigators have found that their patients have regained their range of motion and function earlier and, in some cases, with larger gains compared to their previous patients they had immobilized for 6 weeks before initiating their rehabilitation. The purpose of this study is to compare patients that have been exposed to the early versus standard rehabilitation protocol to see if there is significant improvement in their range of motion, pinch and grip strength, pain levels and function.

ELIGIBILITY:
Inclusion Criteria:

* clinical and radiographic diagnosis of 1st CMC OA
* failed to improve with conservative modalities
* continued pain over the first CMC joint
* loss of strength or motion of the thumb that limits activities of daily living

Exclusion Criteria:

* rheumatoid arthritis
* gout
* cervical radiculopathy
* previous thumb/1st CMC surgery
* post-traumatic arthritis of 1st CMC
* carpal tunnel syndrome with motor function impairment
* patients with post-traumatic arthritis of their 1st CMC AND have dislocation of this joint.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pinch strength | 6 weeks
  standard hydraulic hand dynamometer

SECONDARY OUTCOMES:
range of motion | 6 weeks
  range of hand motion

OTHER OUTCOMES:
Visual analog scale | 6 weeks
  pain measurement
first metacarpal height as measured on xray image | 6 weeks
  measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: David Pichora, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada